CLINICAL TRIAL: NCT02188602
Title: Retrospective Investigation of Chloride Dosing and Its Effect on Acute Kidney Injury
Brief Title: Effect of Cumulative Chloride Dose on Development of Acute Kidney Injury in Critically Ill Children
Status: Withdrawn | Type: Observational
Why Stopped: Researcher left institution
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 27752
Record Dates: First submitted 2013-07-19; First posted 2014-07-11 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High Chloride Dose: Patients receiving high dosing of chloride
- Low Chloride Dose: Patients receiving low dosing of chloride

SUMMARY:
The investigators would like to investigate the effect of chloride dosing on the development of acute kidney injury in critically ill patients. The investigators hypothesis is that administering intravenous fluids with higher chloride content are more likely to lead to acute kidney injury.

DETAILED DESCRIPTION:
Retrospective chart review from 2008-2012 evaluating chloride dosing and serum chloride levels and their effects on acute kidney injury in the pediatric ICU. Patients will be included for the first seven days of their PICU stay.

ELIGIBILITY:
Inclusion Criteria:

* age less than 18 years
* PICU admitting diagnosis of sepsis, respiratory failure, or hepatic failure.

Exclusion Criteria:

* hyponatremia or hypernatremia at PICU admission
* preexisting diagnosis of End-stage renal disease or renal transplant
* presence of neurologic comorbidities.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children < 18 yo admitted to the Pediatric Intensive Care Unit at Lucile Packard Children's Hospital with admitting diagnosis of sepsis, respiratory failure, or liver failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 7 days
  or sooner if death or discharged

SECONDARY OUTCOMES:
PICU length of stay | 7 days
Hospital length of stay | 7 days
Number of ventilator days | 7 days
Mortality | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Weiwen V Shih, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States